CLINICAL TRIAL: NCT04534686
Title: CogXergaming to Promote Physical Activity and Cognitive Function to Enhance Community Mobility and Quality of Life in Frail Older Adults
Brief Title: CogXergaming to Promote Physical Activity and Cognitive Function in Frail Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Tanvi Bhatt, PI, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0280
Record Dates: First submitted 2020-08-27; First posted 2020-09-01 (Actual); Results first posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Frail Older Adults
Keywords: CogXergaming; Dual-task training; Cognitive-motor-balance training
MeSH Terms: interventions — Cognitive Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CogXergaming (Experimental): CogXergaming based cognitive-motor balance training will be delivered to group A using the commercially available Wii-Fit Nintendo and a mouse in conjunction with cognitive training. All participants will undergo 18 sessions of training in a tapering manner for six weeks with 60-90 minutes of training per session, i.e., 3 sessions each week till the 6th week. Each session will be divided into 3 sub-sessions, where each sub-session will consist of playing 4 to 6 games in conjunction with cognitive task. All the games will be performed using a Wii-Fit balance board in front of a TV screen.
  Interventions: Behavioral: CogXergaming
- Matter of Balance Training (Experimental): Participants in group B will undergo matter of balance training for 8 weeks (one session a week for 2 hours/day).
  Interventions: Behavioral: Matter of Balance Training

INTERVENTIONS:
Behavioral: CogXergaming — The participant will play four of the six balance board games Table tilt, Tightrope, Soccer, Balance bubble, Light Run and Basic Step (each game is max 1.5 minutes). Each game will be superimposed with any 3 of the 6 cognitive tasks (word list generation consisting of verbal fluency (VF) and category fluency (CF), digit recall (DR), analogies (AN), mental arithmetic (MA), repeated letter (RL). The cognitive tasks will be randomized making sure that all the cognitive tasks are played with all the games. The cognitive and balance board game scores will be noted on the scoring sheet for each session. A total 10 minutes rest interval between every sub-session will be mandatorily provided.
  Other Names: Cognitive training
  Arms: CogXergaming
Behavioral: Matter of Balance Training — The program emphasizes practical coping strategies that include group discussions, mutual problem solving, exercises to improve strength, coordination and balance, and, a home safety evaluation.
  Other Names: Conventional training
  Arms: Matter of Balance Training

SUMMARY:
Due to the age associated sarcopenia and reduced cardiovascular fitness, frail older adults experience significant decrease in physical function which comprises of mobility, endurance, muscle strength and balance control. The impaired physical function results in poor quality of life and reduced community participation, leading to increased frailty and long-term disability. Further, compared to cognitively intact frail older adults, cognitively impaired frail older adults experience greater deterioration of such physical function, specifically during dual-task performances (i.e., simultaneous performance of cognitive and motor task). This deterioration occurs due to increased cognitive-motor interference as a result of dual-tasking and is known to increase exhaustion among frail older adults. Previous studies have used multicomponent training and have shown to improve physical function and maintain cardiovascular functioning. However, the capacity of such interventions to improve cognitive function along with physical function is not known or unclear. Further, the concurrent comorbidities that occur along with psychosocial issues such as depression present as barriers and lead to reduced compliance to therapy leaving only a few of them to benefit from it. Alternate forms of therapy such as exergaming with explicit cognitive training has shown promising effects in improving motor and motor function in disabled populations. These studies use a cost-effective, off the shelf device such as Nintendo Wii or Microsoft Kinect to deliver the training which is easily available and clinically translatable. Further, such training has demonstrated increase in brain connectivity enhancing cognitive functions associated with balance control. However, there is limited literature examining the effect of exergaming in older frail population and the efficacy of such training is unknown. Therefore, this study proposes a randomized controlled trial to examine the feasibility of CogXergaming program with an aim to improve locomotor-balance control, cognition, muscular system and cardiovascular fitness.

DETAILED DESCRIPTION:
The population of adults aged 60 years and older has been growing with around half of the people older than 85 years estimated to be frail. Age-related changes in multiple systems affecting balance, mobility, muscle strength, motor processing, cognition, nutrition, endurance and physical activity (PA) results in frailty. Studies on frail older adults have reported improvement in mobility and functional level following exercise interventions. Regular physical activity in this population has helped improve cardiovascular conditioning and quality of life, thus allowing these frail older adults a chance at independent living in the community. In addition to physical comorbidities, the presence of psychosocial issues such as depression may act as a barrier to community participation. Several PA interventions have demonstrated limited long-term effect and sustainable behavioral change in this population. An evidence-based fall prevention program called Matter of Balance (MOB) was developed to reduce fall risk and improve physical function and maximize activity participation in older adults. Meanwhile, Exergaming, a task-specific interactive gaming, has been gaining attention as a novel therapeutic alternative that promotes motor recovery in healthy and disabled populations. Exergaming involves repetitive-task specific exercises with movement execution feedback and motivation provided in real time. Studies have shown Exergaming improved symmetrical weight shifting, multi-directional stepping, single-stance, rapid movement training and self-initiated postural weight shifts in the participants. This anticipatory postural control training helps significantly improve balance control and mobility. In addition to the physical function domains that underlie physical frailty, executive cognitive domain functions also predict late-life physiological impairments. Thus, we postulate that PA facilitated through Exergaming and accompanied by simultaneous cognitive training is a novel approach to counter and inhibit frailty associated with physical function and cognitive decline.

Aim 1: To test the feasibility (compliance and effectiveness) of cognitive-motor exergaming (CogXergaming) in the frail older adults and to compare the improvements in behavioral biomarkers in this group across balance, muscle fitness, cardiovascular fitness and global cognition to the group receiving the Matter of Balance training.

Hypothesis: Participants will respond well to CogXergaming training paradigm and demonstrate significant improvements in balance, muscular fitness, cardiovascular fitness and global cognition as compared to the Matter of Balance training group.

Aim 2: To examine the effect of CogXergaming on physical activity levels and quality of life measures post-intervention.

Hypothesis: The participants who received CogXergaming will demonstrate significant improvement in physical activity and quality of life post-training as compared to their own pre-training scores.

Aim 3: To examine the effect of CogXergaming structural and functional connectivity within the cognitive-motor areas pre and post training to establish effect size.

Hypothesis: Post-training, participants will demonstrate improved memory consolidation, attention, motor planning and execution compared to pre-training indicating improved functional connectivity within the cognitive-motor areas.

ELIGIBILITY:
Inclusion Criteria:

1. Older adults aged 60 years or above
2. Walking speed <0.8m/s
3. Self-reported Physical activity <3 hours/week
4. Hand grip strength <30 kgs for men & <20 kgs for women
5. Not on any sedative drugs
6. Can understand & communicate in English
7. Ability to walk more than 30 feet with or without an assistive device

Exclusion Criteria:

1. Participants will not proceed with the study if any of the following occurs at baseline measurement: 1) HR > 85% of age-predicted maximal heart rate (HRmax) (HRmax = 220 - age), 2) systolic blood pressure (SBP) > 165 mmHg and/or diastolic blood pressure (DBP) > 110 mmHg during resting), and/or 3) oxygen saturation (measured by pulse oximeter) during resting < 90%.
2. Unable to stand for 5 minutes without an assistive device (length of a Wii Fit game)
3. Uncontrolled acute medical/surgical, neurological or cardiovascular disease
4. History of bone fracture or significant other systemic disease or surgery in the last six months
5. Moderate to severe cognitive impairment (MOCA <24/30)
6. Specific to MRI participants: Self-reported presence of pacemaker, metal implants other than orthopedic implants, and/or Claustrophobia, cataract surgery (lens not compatible to the MRI confirmed by the MRI technician)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2021-01-10 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2023-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tanvi S Bhatt, PT,MS,PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Kannan L, Sahu U, Subramaniam S, Mehta N, Kaur T, Hughes S, Bhatt T. Gaming-Based Tele-Exercise Program to Improve Physical Function in Frail Older Adults: Feasibility Randomized Controlled Trial. J Med Internet Res. 2024 Nov 27;26:e56810. doi: 10.2196/56810. PMID 39602215

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We initially recruited the participants by posting flyers (approved by the Institutional Review Board) at Geriatric and internal medicine by contacting collaborators, giving presentations to potential participants at various exercise centers and senior homes. We will also use social media, such as Facebook, Twitter, etc. to post flyer for recruitment
Period: Baseline Measurement
Arm/Group | CogXergaming | Matter of Balance Training
Started | 22 | 23
Mid-intervention | 18 | 18
Completed | 15 | 16
Not Completed | 7 | 7
Not completed — Lost to Follow-up | 4 | 6
Not completed — Withdrawal by Subject | 3 | 1
Period: Intervention
Arm/Group | CogXergaming | Matter of Balance Training
Started | 15 | 16
Completed | 13 | 14
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CogXergaming | Matter of Balance Training | Total
Number analyzed (Participants) | 22 | 23 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.15 (6.03) | 71.83 (5.98) | 72.13 (5.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 30
  Male | 6 | 9 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 4 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 8 | 18
  White | 8 | 11 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Montreal Cognitive Assessment [Mean (Standard Deviation); unit: units on a scale] — The Montreal Cognitive Assessment is a scoring system used to assess cognitive function. The minimum possible score of the assessment is 0 points and the maximum possible score is 30 points. Higher score indicates better performance. A score of above 24 points indicates intact cognition.
  units on a scale | 27.34 (5.01) | 27.60 (4.82) | 27.36 (4.82)

OUTCOME MEASURES:

1. Primary Outcome: Change in 30-second Chair Stand Performance
Description: This test is conducted to assess leg strength and endurance. Participants are asked to stand in front of a sturdy chair and monitored by the remote research personnel during the test. The participants are instructed to sit in the middle of the chair. Place their hands on the opposite shoulder crossed, at the wrists. Keep their feet flat on the floor and back straight with arms against their chest. Then the following instruction "On "Go," rise to a full standing position, then sit back down again. 6. Repeat this for 30 seconds" is provided to conduct the test and assessed by the research personnel remotely. This test is easy to perform and requires a sturdy chair (available at every home) and will be performed in front of the camera during the zoom meeting for the research personnel to monitor and collect the required data. Higher values indicate better performance
Time Frame: Baseline (Week 0) and Immediate Post-training (Week 8 for group A and week 10 for group B)
Population: 13 participants in the Coxergaming and 14 in the Matter of Balance group completed the study and data was analyzed for these participants.
Measure: Mean (Standard Deviation); unit: number of repetitions
Arm/Group | CogXergaming | Matter of Balance Training
Number analyzed (Participants) | 13 | 14
number of repetitions
  Baseline | 10.28 (1.63) | 12.11 (1.81)
  Immediate Post-training | 12.36 (1.62) | 12.30 (1.53)

2. Primary Outcome: Change in Walking Performance
Description: Walking performance will be assessed using the Tinetti Performance Oriented Mobility Assessment. This test contains components of gait and balance assessment and is scored on a scale, typically from 0 to 2, with higher scores indicating better performance. The total score combines the scores from both sections, with a minimum score of 0 and a maximum score of 28. This test will be evaluated remotely over zoom. A safe area visible to the research personnel remotely will be chosen and only then the test will be administered. During this test, the research personnel will ensure that he/she is constantly visible in the screen and measure the time taken to complete the test. Higher scores on the test indicate better performance.
Time Frame: Baseline (Week 0) and Immediate Post-training (Week 8 for group A and week 10 for group B)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale of 28
Arm/Group | CogXergaming | Matter of Balance Training
Number analyzed (Participants) | 13 | 14
scores on a scale of 28
  Baseline | 25.93 (2.12) | 26.95 (1.16)
  Immediate Post-training | 26.92 (0.75) | 26.93 (1.22)

3. Primary Outcome: Change in Cardiovascular Fitness
Description: Cardiovascular fitness will be assessed using the 2-min step test, which will be conducted remotely via zoom. The participant is asked to stand up straight next to the wall while a mark is placed on the wall at the level corresponding to midway between the kneecap and top of the hip bone. The subject then marches in place for two minutes, lifting the knees to the height of the mark on the wall. Resting is allowed and holding onto the wall or a stable chair is allowed. Stop after two minutes of stepping. The remote research personnel records the total number of times the right knee reaches the tape level in two minutes. Higher scores on the test indicate better performance
Time Frame: Baseline (Week 0) and Immediate Post-training (Week 8 for group A and week 10 for group B)
Measure: Mean (Standard Deviation); unit: number of repetitions
Arm/Group | CogXergaming | Matter of Balance Training
Number analyzed (Participants) | 13 | 14
number of repetitions
  Baseline | 75.06 (16.51) | 78.61 (10.97)
  Immediate Post-training | 85.45 (11.52) | 82.71 (10.27)

4. Primary Outcome: Change in Physical Activity
Description: Physical activity will be assessed remotely via zoom using the scoring of the Physical Activity Scale for the Elderly (PASE) involves assigning weights to different types of physical activities based on their intensity and frequency. Respondents report their weekly frequency and duration of various activities, which are then multiplied by predetermined weights. The total PASE score is the sum of these weighted values, providing a single numeric value representing the individual's overall physical activity level. Higher scores indicate higher levels of physical activity. The minimum score for PASE is 0 and maximum score is 793.
Time Frame: Baseline (Week 0) and Immediate Post-training (Week 8 for group A and week 10 for group B)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale of 793
Arm/Group | CogXergaming | Matter of Balance Training
Number analyzed (Participants) | 13 | 14
scores on a scale of 793
  Baseline | 72.68 (38.10) | 77.11 (40.8)
  Immediate post-training | 110.03 (23.80) | 92.49 (29.4)

5. Primary Outcome: Change in Movement Velocity
Description: It is the average speed of center of gravity movement during intentional movement measured in degrees per second under single and dual-task conditions. Higher values indicate better performance.
Time Frame: Baseline (Week 0) and Immediate Post-training (Week 8 for group A and week 10 for group B)
Population: Due to the emergence of the COVID-19 pandemic, this study was conducted primarily on Zoom, preventing the collection of data for this outcome measure, as the assessment is typically conducted in person.
Arm/Group | CogXergaming | Matter of Balance Training
Number analyzed (Participants) | 0 | 0

6. Primary Outcome: Change in End Point Excursion
Description: It is the magnitude of a self-initiated movement (i.e., how far he/she wills to reach a target) without taking a step or losing balance measured in percentage under single and dual-task conditions. Higher values indicate better performance.
Time Frame: Baseline (Week 0) and Immediate Post-training (Week 8 for group A and week 10 for group B)
Population: as for outcome 5
Arm/Group | CogXergaming | Matter of Balance Training
Number analyzed (Participants) | 0 | 0

7. Primary Outcome: Change in Directional Control
Description: It is the quality of a self-initiated movement (i.e., amount of movement actually exhibited towards the target to the amount of extraneous movement away from the target) measured in percentage under single and dual-task conditions. Higher values indicate better performance.
Time Frame: Baseline (Week 0) and Immediate Post-training (Week 8 for group A and week 10 for group B)
Population: as for outcome 5
Arm/Group | CogXergaming | Matter of Balance Training
Number analyzed (Participants) | 0 | 0

8. Primary Outcome: Change in Maximum Excursion
Description: It is the actual magnitude of a self-initiated movement (i.e., how far did he/she actually reach a target) without taking a step or losing balance measured in percentage under single and dual-task conditions. Higher values indicate better performance.
Time Frame: Baseline (Week 0) and Immediate Post-training (Week 8 for group A and week 10 for group B)
Population: as for outcome 5
Arm/Group | CogXergaming | Matter of Balance Training
Number analyzed (Participants) | 0 | 0

9. Primary Outcome: Change in Postural Stability During Reactive Balance Control (Single and Dual-task)
Description: Reactive balance control will be examined via the stance perturbation test under single and dual-task conditions (simultaneous performance of Letter number sequencing task or auditory stroop task). Postural stability can be defined as simultaneous control of center of mass (COM) position and velocity during slip-like or trip like perturbation relative to the rear edge of base of support (rear heel). The position is normalized with the individual's foot length, and velocity by square root of gravitational acceleration and individual's body height. Larger values indicate greater stability.
Time Frame: Baseline (Week 0) and Immediate Post-training (Week 8 for group A and week 10 for group B)
Population: as for outcome 5
Arm/Group | CogXergaming | Matter of Balance Training
Number analyzed (Participants) | 0 | 0

10. Primary Outcome: Change of Accuracy in Letter Number Sequencing
Description: This is an oral trail making test which includes listing alternate letter and number from the cue given in sequence. This test will be performed under single and dual-task conditions.
  Accuracy (number of correct responses out of the total responses) of letter number sequencing will be calculated. Higher accuracy indicates better performance.
Time Frame: Baseline (Week 0) and Immediate Post-training (Week 8 for group A and week 10 for group B)
Population: as for outcome 5
Arm/Group | CogXergaming | Matter of Balance Training
Number analyzed (Participants) | 0 | 0

11. Primary Outcome: Change in 4 Meter Walk Test
Description: The total time taken to complete the 4 meters will be noted. Speed will then be determined by using the formula distance (4 meters) covered by time taken to complete the test. Higher speed indicates better performance.
Time Frame: Baseline (Week 0) and Immediate Post-training (Week 8 for group A and week 10 for group B)
Population: as for outcome 5
Arm/Group | CogXergaming | Matter of Balance Training
Number analyzed (Participants) | 0 | 0

12. Primary Outcome: Change in Spatial and Temporal Gait Parameters
Description: Spatial and temporal gait parameters like step length, cadence and stride length will be determined during single and dual-task walking performance via the GaitRite mat. Higher values for step length and stride length, and lower cadence indicates better performance.
Time Frame: Baseline (Week 0) and Immediate Post-training (Week 8 for group A and week 10 for group B)
Population: as for outcome 5
Arm/Group | CogXergaming | Matter of Balance Training
Number analyzed (Participants) | 0 | 0

13. Primary Outcome: Change in Accuracy of Auditory Stroop
Description: This test involves responding to the pitch (high or low) of the words "High" or "Low". This test will be performed under single and dual-task conditions.
  Accuracy (number of correct responses out of the total responses) of Auditory stroop will be calculated. Higher accuracy indicates better performance. Higher values indicate better performance.
Time Frame: Baseline (Week 0) and Immediate Post-training (Week 8 for group A and week 10 for group B)
Population: as for outcome 5
Arm/Group | CogXergaming | Matter of Balance Training
Number analyzed (Participants) | 0 | 0

14. Primary Outcome: Change in Dual-task Cost
Description: Dual-task motor and cognitive cost will be calculated using the formula- [(Dual-task performance- Single Task performance)/Single task performance]. This will be calculated for dual-task performance during intentional postural sway, reactive balance control and gait conditions. Lower cost indicates better performance.
Time Frame: Baseline (Week 0) and Immediate Post-training (Week 8 for group A and week 10 for group B)
Population: as for outcome 5
Arm/Group | CogXergaming | Matter of Balance Training
Number analyzed (Participants) | 0 | 0

15. Primary Outcome: Change in Interference in the Reaction Time
Description: Interference in the reaction time via visual stroop task where the individual is expected to respond to the color in which the word is printed and not read the word. Performance will be identified via time taken to complete the test. Lower time indicates better performance.
Time Frame: Baseline (Week 0) and Immediate Post-training (Week 8 for group A and week 10 for group B)
Population: as for outcome 5
Arm/Group | CogXergaming | Matter of Balance Training
Number analyzed (Participants) | 0 | 0

16. Primary Outcome: Change in Language Fluency
Description: Language fluency via verbal and category task will be administered. Performance will be identified via the total number of appropriate words responded on each of the task. Higher values indicate better performance.
Time Frame: Baseline (Week 0) and Immediate Post-training (Week 8 for group A and week 10 for group B)
Population: as for outcome 5
Arm/Group | CogXergaming | Matter of Balance Training
Number analyzed (Participants) | 0 | 0

17. Primary Outcome: Change in Reaction Time
Description: The individual is asked to hit a key on the number keypad when a cue appears on the screen. Performance will be identified with time taken to hit the key after the individual sees the cue in seconds. Lower time indicates better performance.
Time Frame: Baseline (Week 0) and Immediate Post-training (Week 8 for group A and week 10 for group B)
Population: as for outcome 5
Arm/Group | CogXergaming | Matter of Balance Training
Number analyzed (Participants) | 0 | 0

18. Primary Outcome: Change in Paired Associated Learning
Description: Paired associated learning via grid task will be administered. Accuracy (number of correct responses out of the total responses) will be represented in percentage. Higher value indicates better performance.
Time Frame: Baseline (Week 0) and Immediate Post-training (Week 8 for group A and week 10 for group B)
Population: as for outcome 5
Arm/Group | CogXergaming | Matter of Balance Training
Number analyzed (Participants) | 0 | 0

19. Primary Outcome: Change in Spatial Working Memory
Description: Spatial working memory via unveil the star task will be administered. Performance will be identified via the total time (in seconds) to complete the task. Lower time indicates better performance.
Time Frame: Baseline (Week 0) and Immediate Post-training (Week 8 for group A and week 10 for group B)
Population: as for outcome 5
Arm/Group | CogXergaming | Matter of Balance Training
Number analyzed (Participants) | 0 | 0

20. Primary Outcome: Change in Working Memory
Description: List Sorting Memory test to evaluate working memory. This test requires the participant to recall and sequentially list the visually and orally presented stimuli. The accuracy of the participant's response is computer generated. Higher value indicates better performance. The minimum score is 0% and maximum score is 100%
Time Frame: Baseline (Week 0) and Immediate Post-training (Week 8 for group A and week 10 for group B)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | CogXergaming | Matter of Balance Training
Number analyzed (Participants) | 13 | 14
percentage
  Baseline | 16.11 (3.3) | 16.22 (3.3)
  Immediate post-training | 16.85 (3.93) | 16.11 (2.93)

21. Primary Outcome: Change in Episodic Memory
Description: Picture sequence memory test will assess episodic memory of the individual. The number of adjacent pairs of pictures placed correctly will score a point. The scores are computer generated. Higher value indicates better performance.
Time Frame: Baseline (Week 0) and Immediate Post-training (Week 8 for group A and week 10 for group B)
Population: as for outcome 5
Arm/Group | CogXergaming | Matter of Balance Training
Number analyzed (Participants) | 0 | 0

22. Primary Outcome: Change in Accuracy of Flanker Inhibitory Control and Attention Test
Description: Flanker inhibitory control and attention test is used to evaluate the participant's ability to inhibit the attention to the stimulus flanking it and focus on a particular stimulus. Accuracy of the responses are recorded and the scores are computer generated. Higher value indicates better performance.
Time Frame: Baseline (Week 0) and Immediate Post-training (Week 8 for group A and week 10 for group B)
Population: as for outcome 5
Arm/Group | CogXergaming | Matter of Balance Training
Number analyzed (Participants) | 0 | 0

23. Primary Outcome: Change in Cognitive Flexibility and Attention
Description: Dimensional Change card sort assesses cognitive flexibility and attention. Participants are asked to match a series of bivalent pictures either by colors or shapes accordingly. Responses are computer recorded and accuracy scores are computer generated. Higher value indicates better performance.
Time Frame: Baseline (Week 0) and Immediate Post-training (Week 8 for group A and week 10 for group B)
Population: as for outcome 5
Arm/Group | CogXergaming | Matter of Balance Training
Number analyzed (Participants) | 0 | 0

24. Primary Outcome: Change in Processing Speed
Description: Pattern comparison processing speed test is used to evaluate the processing speed. The participants are expected to respond whether the two pictures side-by side are same or not the same. Accuracy will be recorded by the computer and scores are computer generated. Higher value indicates better performance.
Time Frame: Baseline (Week 0) and Immediate Post-training (Week 8 for group A and week 10 for group B)
Population: as for outcome 5
Arm/Group | CogXergaming | Matter of Balance Training
Number analyzed (Participants) | 0 | 0

25. Primary Outcome: Changes in Fractional Anisotropy
Description: Image acquisition will be performed in a 3T and 1.5T Magnetic resonance scanner (MR 750, GE healthcare, Milwaukee). Fractional anisotropy (FA) is a scalar value ranging from 0-1 and change from pre- to post-training will compared to determine the structural and functional connectivity. Increase in FA values post-training will indicate positive results of training.
Time Frame: Baseline (Week 0) and Immediate Post-training (Week 8 for group A and week 10 for group B)
Population: as for outcome 5
Arm/Group | CogXergaming | Matter of Balance Training
Number analyzed (Participants) | 0 | 0

26. Secondary Outcome: Berg Balance Scale
Description: Assess static and dynamic balance. This scale consists of the participant transferring from one chair to another, reaching forward, stepping up and down from a stepping stool, standing with eyes closed and open, one leg standing. It is a 14-item scale with each item score ranging from 0-4. Performance on the scale will be calculated on a total of 56. Less than 45 will indicate greater risk of falling.
Time Frame: Baseline (Week 0) and Immediate Post-training (Week 8 for group A and week 10 for group B)
Population: as for outcome 5
Arm/Group | CogXergaming | Matter of Balance Training
Number analyzed (Participants) | 0 | 0

27. Secondary Outcome: Change in Physical Activity Level (Questionnaires)
Description: Questionnaires such as Physical Activity Scale for elderly and activity specific balance confidence scale will be self-reported by the participant. Activity specific balance confidence scale consists of 16 items, and each item score ranges from 0-100. The total score with 0 confidence indicates no confidence and 100 with complete confidence.
Time Frame: Baseline (Week 0) and Immediate Post-training (Week 8 for group A and week 10 for group B)
Population: as for outcome 5
Arm/Group | CogXergaming | Matter of Balance Training
Number analyzed (Participants) | 0 | 0

28. Secondary Outcome: Change in Physical Activity Level
Description: Average number of steps taken a day by the individual prior to and after training.
Time Frame: Baseline (Week 0) and Immediate Post-training (Week 8 for group A and week 10 for group B)
Population: as for outcome 5
Arm/Group | CogXergaming | Matter of Balance Training
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline through study completion, which includes 8 weeks for Cogxergaming and 10 weeks for Matter of Balance
Arm/Group | CogXergaming | Matter of Balance Training
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/23
Other Adverse Events (participants affected / at risk) | 0/22 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-26): https://cdn.clinicaltrials.gov/large-docs/86/NCT04534686/Prot_SAP_000.pdf